CLINICAL TRIAL: NCT03422432
Title: Pilot Study: Prophylactic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Colorectal Cancers at High Risk of Developing Peritoneal Metastases
Brief Title: Prophylactic HIPEC for Colorectal Cancers at High Risk of Developing Peritoneal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/2402/B
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Patients are identified pre-operatively on radiological imaging. Prophylactic HIPEC will be delivered intra-operatively, immediately after the resection of the primary tumour, and only if the patient is deemed well enough to receive the HIPEC.
  Interventions: Procedure: HIPEC
- Group 2 (Experimental): Patients are identified post-operative based on histological findings. They will be counselled to receive prophylactic HIPEC only. If peritoneal nodules are found during surgery, these patients will be excluded from the study.
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — All HIPEC will be with Mitomycin C and given at a dose of 10mg/body surface area.

SUMMARY:
The study investigators hypothesize that prophylactic HIPEC is feasible and well tolerated in patients with colorectal cancers with high-risk of developing peritoneal recurrence.

The aim of the pilot study is to test the feasibility of performing prophylactic HIPEC for colorectal cancer patients at high-risk of developing peritoneal recurrence in our institution, and determine the morbidity associated with such a procedure.

Patients with high-risk of developing peritoneal recurrence are defined as patients with

1. tumours involving the serosa and adjacent viscera (i.e. T4 cancers)
2. krukenburg tumours (i.e. ovarian metastases)
3. perforated tumours
4. positive peritoneal fluid cytology
5. minimal synchronous PC (nodules <1cm in the omentum and/or close to the primary tumour).

The study investigators plan to assess feasibility according to

1. The number of patients completing the treatment
2. Time to adjuvant systemic chemotherapy, to evaluate if there is delay to adjuvant treatment

Morbidity will be measured according to the Clavien-Dindo Classification, and graded according to low versus high grade morbidity.

If prophylactic HIPEC is shown to be feasible, with acceptable morbidity, the investigators aim to carry out a randomized controlled trial to determine the effectiveness of prophylactic HIPEC in preventing the development of peritoneal metastases in patients with colorectal cancer at high risk of peritoneal recurrence.

ELIGIBILITY:
Inclusion Criteria:

Two groups of patients may be enrolled:

Group 1 patients are identified pre-operatively on radiological imaging, while Group 2 patients are identified post-operative based on histological findings.

All patients diagnosed with adenocarcinoma of the colon and rectum, and either one of the five following risk factors for peritoneal metastases will be considered for inclusion:

1. T4 tumours - in Group 1, this would consist of obvious clinical T4 stage based on preoperative imaging, and in Group 2, this would be on pathological confirmation of a T4 tumour.
2. Krukenburg tumours - Unilateral or bilateral ovarian masses seen on preoperative imaging
3. Perforated tumours - in Group 1, this would consist of patients presenting with perforation on preoperative imaging, and undergoing curative resection, and in Group 2, this would be on pathological or intra-operative confirmation of a perforated tumour.
4. Limited synchronous peritoneal metastases (peritoneal nodules <1cm in the omentum and/or close to the tumour). Patients with limited peritoneal disease in close proximity to the primary tumour, that may be removed enbloc with the primary resection can be included, but patients with more extensive peritoneal disease and those with extra-peritoneal metastases i.e. liver and/or lung metastases will be excluded from the study.
5. Positive cytology in Group 2 patients

Other inclusion criteria:

1. Patients must be between the ages of 21 and 75 years
2. Patients must be in a stable clinical condition to undergo simultaneous HIPEC after the primary curative colorectal resection
3. Patients must have an ECOG performance status 0 or 1
4. Patients must have normal organ and marrow function as defined below:

i. Absolute neutrophil count > 1.5 x 109/L ii. Platelets > 100 x 109/L iii. Haemoglobin > 9.0g/dl iv. Total bilirubin ≤1.5 x ULN v. AST(SGOT)/ALT(SGPT) < 3 X institutional ULN vi. Creatinine ≤1.5 x upper limit of normal (ULN) OR vii. Creatinine clearance ≥60 mL/min for patients with creatinine levels >1.5 x institutional UL e. Patients must have a normal coagulation profile f. Patients must give written informed consent

Exclusion Criteria:

1. Patients who are not fit to give consent for the procedure
2. Patients who are not fit to undergo surgery
3. Patients who are pregnant
4. Patients who have extensive synchronous peritoneal disease
5. Patients with extra-peritoneal metastases i.e. liver and/or lung metastases

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
The number of patients completing the treatment | From start to end of study, approximately 1 year
Time to adjuvant systemic chemotherapy | 3 months from date of surgery
  To evaluate if there is delay to adjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Grace Tan, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No